CLINICAL TRIAL: NCT03142061
Title: Prospective Evaluation of Clinical Efficacy and Symptom Control Using Electrochemotherapy for the Inoperable Advanced Vulva Carcinoma
Brief Title: Electrochemotherapy for the Inoperable Vulva Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 558/2015BO1
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2020-02

CONDITIONS: Advanced Inoperable Vulva Carcinoma
MeSH Terms: interventions — Electrochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECT (Experimental)
  Interventions: Procedure: Electrochemotherapy

INTERVENTIONS:
Procedure: Electrochemotherapy — Bleomycin plus local electroporation of cutan accessible tumor tissue in patients with advanced inoperable vulva carcinoma

SUMMARY:
Electrochemotherapy (ECT) with Bleomycin in non-operable advanced vulva carcinoma

DETAILED DESCRIPTION:
Prospective evaluation of tumor response towards ECT by photo documentation. In addition prospective documentation of life quality after ECT treatment as well as evaluation of pain. .

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age ≥ 55 years (postmenopausal)
* histologically proved cutan accessible vulva carcinoma
* a maximum of 5 lesions ≥1 - ≤ 5 cm diameter; a maximum thickness of 3 cm
* applied electrochemotherapy with electroporation

Exclusion Criteria:

* Non compliant patients
* Patients with symptomatic or rapidly progredient metastasis outside of the vulva

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
local tumor control | Baseline
  according to RECIST criteria
Symptom control | Baseline
  exulceration, secretion

SECONDARY OUTCOMES:
Life quality | Baseline, 3, 6 months
  EORTC QLQ
Pain | Baseline, 3, 6 months
  Visual scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No